CLINICAL TRIAL: NCT01540422
Title: OPTION Trial: Optimal Improvement of Vein Graft Patency Long Term by the Implementation Of Novel Endoscopic Harvesting Techniques
Brief Title: Study to Improve Long Term Vein Graft Patency After Coronary Bypass Surgery by Using a Novel Endoscopic Harvesting Technique
Status: Completed | Type: Observational
Sponsor: Baylor Research Institute (Other)
Collaborators: Maquet Cardiovascular (Industry)
Responsible Party: Sponsor
Other Study IDs: 009-177
Record Dates: First submitted 2012-02-23; First posted 2012-02-28 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2015-03

CONDITIONS: Coronary Artery Disease
Keywords: vein grafts; coronary bypass; endoscopic harvest; endoscopic vein harvest
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- CABG w/saphenous vein grafts harvested using endoscopy: Those who have CABG surgery with saphenous vein grafts harvested using endoscopic techniques

SUMMARY:
The purpose of this study is to demonstrate improved vein graft patency rates at 12 months for endoscopically harvested saphenous vein grafts. The study will evaluate use modifications to existing techniques in vein graft handling during harvests. A secondary aim is to develop a standardized approach for harvesting, handling, and preparing vein grafts in the endoscopic approach.

DETAILED DESCRIPTION:
Available data supports two facts: 1) Saphenous vein graft failure rates may be as high as 47% per patient at one year post coronary artery bypass grafting, and 2) Endoscopic vein-graft harvesting is independently associated with vein-graft failure and adverse clinical outcomes.

Multiple factors may contribute to the lower long term patency rates of endoscopically harvested grafts. Summarized, the two major contributing factors are theorized to be harvesting techniques and vein trauma during harvesting.

With recognized disadvantages of open vessel harvesting including higher incidence of infection, longer incisions, greater potential for poor healing, and longer length of hospital stay, reducing the failure rate of vein grafts harvested endoscopically is of utmost importance.

It is our hypothesis that modification of existing harvesting techniques can improve vein graft patency in endoscopic vein graft harvesting so that patency rates comparable to open vessel harvesting can be obtained.

In this prospective, multi-center non-randomized, observational study, 100 patients will undergo routine coronary artery bypass grafting. Eligible candidates will undergo lone coronary artery bypass graft (CABG) procedures with endoscopic vein graft harvesting using best harvesting practices. As a part of routine postoperative care, patients will be prescribed dual-antiplatelet therapy of aspirin and clopidogrel. Compliance with 3 months of dual-antiplatelet therapy will be monitored.

Vein graft patency will be evaluated:

1. Intra-operatively by transit time graft flow measurements.
2. Post-operative Day 30 through Cardiac CT Angiography.
3. Post-operative Month 12 through Cardiac CT Angiography.

ELIGIBILITY:
Inclusion Criteria:

* Males and females at least 18 years of age and able to sign consent
* Undergoing CABG surgery
* Eligible for endoscopic saphenous vein harvesting
* A minimum of two non-sequential vein grafts will be performed
* Subject willing to comply with the requirements of the protocol

Exclusion Criteria:

1. Previous CABG
2. Previous or concomitant valve surgery
3. Any other concomitant cardiac procedure other than surgical ablation or incidental PFO repair
4. Intolerance to Iodine or IV contrast that cannot be controlled with pre-medication
5. Renal insufficiency with GFR measurement ≤ 40, unless dialysis dependent
6. Abnormal platelet level defined as Plt Count >400,000
7. Abnormal platelet function (hypercoagulable state) as evidenced by TEG testing
8. Allergy to or presence of a condition that the investigator feels may prevent safe administration of ASA or Plavix post-operatively.
9. Patient has a co-morbid condition that in the opinion of the investigator poses undue risk for successful endovascular harvesting of the vein

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospital facility
Sampling Method: Non-Probability Sample
Enrollment: 93 (Actual)
Dates: Start 2010-10; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Improved vein graft patency | Baseline and 12 months
  To demonstrate improved vein graft patency at 12 months for endoscopically harvested saphenous vein grafts by using modifications to existing vein harvest techniques in vein handling during harvest.

SECONDARY OUTCOMES:
Vein graft failure | Baseline, 30 days, and 12 months
  1. Assess the incidence of vein graft failure at the time of initial CABG as evaluated by transit time graft flow measurements.
  2. Incidence of vein graft failure at postoperative day 30 as evaluated by Coronary CT angiography
  3. Incidence of vein graft failure at postoperative Month 12 as evaluated by Coronary CT angiography
  4. Incidence of vein graft failure at each interval (30 day and 12 month) as categorized by:
     1. Harvested vessel (greater versus lesser saphenous vein)
     2. Vein graft destinations
     3. Vein graft quality

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Medical City Hospital, Dallas, Texas
  - The Heart Hospital Baylor Plano, Plano, Texas

REFERENCES:
- [Background] Bolotin G, Kypson AP, Nifong LW, Chitwood WR Jr. A technique for evaluating competitive flow for intraoperative decision making in coronary artery surgery. Ann Thorac Surg. 2003 Dec;76(6):2118-20. doi: 10.1016/s0003-4975(03)00652-0. PMID 14667667
- [Result] Lopes RD, Hafley GE, Allen KB, Ferguson TB, Peterson ED, Harrington RA, Mehta RH, Gibson CM, Mack MJ, Kouchoukos NT, Califf RM, Alexander JH. Endoscopic versus open vein-graft harvesting in coronary-artery bypass surgery. N Engl J Med. 2009 Jul 16;361(3):235-44. doi: 10.1056/NEJMoa0900708. PMID 19605828
- [Result] Burris N, Schwartz K, Tang CM, Jafri MS, Schmitt J, Kwon MH, Toshinaga O, Gu J, Brown J, Brown E, Pierson R 3rd, Poston R. Catheter-based infrared light scanner as a tool to assess conduit quality in coronary artery bypass surgery. J Thorac Cardiovasc Surg. 2007 Feb;133(2):419-27. doi: 10.1016/j.jtcvs.2006.09.056. Epub 2006 Dec 29. PMID 17258576
- [Result] Serruys PW, Morice MC, Kappetein AP, Colombo A, Holmes DR, Mack MJ, Stahle E, Feldman TE, van den Brand M, Bass EJ, Van Dyck N, Leadley K, Dawkins KD, Mohr FW; SYNTAX Investigators. Percutaneous coronary intervention versus coronary-artery bypass grafting for severe coronary artery disease. N Engl J Med. 2009 Mar 5;360(10):961-72. doi: 10.1056/NEJMoa0804626. Epub 2009 Feb 18. PMID 19228612